CLINICAL TRIAL: NCT04791397
Title: Double-Blind, Placebo-Controlled, Randomized Parallel Design Trial of Evaluation of the Effect of Interval Hypoxic-hyperoxic Training (IHHT) on Vascular Stiffness and Elasticity of the Liver Tissue in Patients With Metabolic Syndrome.
Brief Title: Evaluation of the Effect of IHHT on Vascular Stiffness and Elasticity of the Liver Tissue in Patients With MS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0519
Record Dates: First submitted 2020-05-13; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-05

CONDITIONS: Vascular Stiffness; Liver Fibroses; Metabolic Syndrome; Trimethylamine N-oxyde; Toll-like Receptors
Keywords: Metabolic syndrome; Vascular Aging; Non-alcoholic Fatty Liver Disease; Non-drug methods; Interval Hypoxic-hyperoxic training; Trimethylamine N-oxyde (TMAO); Toll-like Receptors (TLR)
MeSH Terms: conditions — Liver Cirrhosis; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group trial (Experimental): Included 30 patients, with metabolic syndrome, aged 24-71 year old.
  Interventions: Procedure: Interval hypoxic-hyperoxic training (IHHT) using respiratory therapy unit ReOxy.
- Group control (Experimental): Included 30 patients, with metabolic syndrome, aged 24-71 year old.
  Interventions: Procedure: Simulating Interval hypoxic-hyperoxic training (IHHT) using respiratory therapy unit ReOxy.

INTERVENTIONS:
Procedure: Interval hypoxic-hyperoxic training (IHHT) using respiratory therapy unit ReOxy. — Every patient from control group undergo 15 procedures of IHHT, 5 procedures per week for 3 weeks, 1 procedure lasts 40 minutes. IHHT is a protocol which employs passive (the patient is at rest), short (several minutes) mild normobaric hypoxic exposures alternated with similar duration intervals of breathing hyperoxia, and repeated for 40 minutes. During the initial pretreatment test, the patient inhales air with low oxygen content at atmospheric pressure in a continuous mode through a mask. In the interval therapeutic mode that follows, periods of hypoxia (10-14% O2) are interrupted by periods of reoxygenation by hyperoxia (up to 35% O2). Automatic switching of gas flows (SRT technology). Built-in intelligent software automatically identifies and suggests key treatment parameters for the individual treatment program, by adjusting the starting parameters based upon the results of the pretreatment hypoxic test.
  Arms: Group trial
Procedure: Simulating Interval hypoxic-hyperoxic training (IHHT) using respiratory therapy unit ReOxy. — Every patient from group control undergo simulating procedures of interval hypoxic-hyperoxic training, 15 procedures, 5 procedures per week for 3 weeks. 1 procedure lasts 40 minutes, in normoxia. Before the start of the course, each patient undergoes a test procedure for 10 minute (in normoxia) for simulate procedures IHHT.
  Arms: Group control

SUMMARY:
The aim of this study is to assess the effect of interval hypoxy-hyperoxic training (IHHT) on the arterial stiffness and elasticity of the liver tissue in patients with metabolic syndrome and on other components of the metabolic syndrome, and the possibility of their reversible recovery after training.

DETAILED DESCRIPTION:
The study will included 60 patients with metabolic syndrome (alimentary obesity (large waist, that measures at least 89 centimeters for women, and 102 centimeters for men), high blood pressure (130/85 mm Hg or higher), dislipidemia (triglyceride level 150 mg/dL (1.7 mmol/L) or higher of this type of fat found in blood; reduced high-density lipoprotein (HDL) cholesterol less than 40 mg/dL (1.04 mmol/L) in men, or less than 50 mg/dL (1.3 mmol/L) in women of HDL cholesterol), elevated fasting blood sugar (100 mg/dL (5,6 mmol/L) or higher). All patients were random separated into two groups: trial (30 pers., who will undergo 15 procedures of the IHHT, 5 days a week for 3 weeks), and control (30 pers., who will undergo 15 placebo procedures simulating IHHT, 5 days a week for 3 weeks). Before and after procedures of IHHT all patients will undergo laboratory and instrumental examinations, wich include arterial stiffness measurement, making by Fukuda Denshi VS-100 VaSera, measurement of liver tissue elasticity and fibrosis, making by elastography on FibroScan (Echosense, XL-sensor), and laboratory analysis (lipid profile, fasting blood sugar, trimethylamin N-oxyde (TMAO), Toll-like receptors 4,7,9). After 6 month of IHHT all patients will undergo the same laboratory and instrumental examinations to assess the duration of the effect.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent.
* The presence of metabolic syndrome: as having three or more of the following traits, including traits you're taking medication to control:
* Large waist - A waistline that measures at least 35 inches (89 centimeters) for women and 40 inches (102 centimeters) for men;
* High triglyceride level - 150 milligrams per deciliter (mg/dL), or 1.7 millimoles per liter (mmol/L), or higher of this type of fat found in blood;
* Reduced "good" or HDL cholesterol - Less than 40 mg/dL (1.04 mmol/L) in men or less than 50 mg/dL (1.3 mmol/L) in women of high-density lipoprotein (HDL) cholesterol;
* Increased blood pressure - 130/85 millimeters of mercury (mm Hg) or higher;
* Elevated fasting blood sugar - 100 mg/dL (5.6 mmol/L) or higher.
* Must be able to come to the hospital 5 days per week, for 3 weeks.

Exclusion Criteria:

* Refusal from further participation in the study.
* Individual intolerance to hypoxia.
* Cirrhosis of the liver with liver failure class C according to the classification of Child-Pugh.
* Alcohol use 140 g / week or more for men, and 70 g / week or more for women.
* Patients with positive serological reactions to hepatitis B and C.
* Chronic kidney disease (GFR less than 30 ml / min / 1.73 m 2).
* Pregnancy, lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Assess the effect of interval hypoxy-hyperoxic training (IHHT) on the arterial stiffness. | Assessment will be measured next day after 15th procedure of the IHHT procedure.
  Assessment of arterial stiffness will be measured by pulse wave velocity using VASERA VS-1500 Fukuda Denshi on next day after course of 15 procedures of IHHT.
Assess the effect of interval hypoxy-hyperoxic training (IHHT) on the liver fibrosis. | Assessment will be measured next day after 15th procedure of the IHHT procedure.
  Assessment of the liver fibrosis and elasticity of liver tissue will be measurement by elastography on FibroScan (Echosense, XL-sensor) by measured liver tissue stiffness (in KPa).

SECONDARY OUTCOMES:
Assess the effect of interval hypoxy-hyperoxic training (IHHT) on the lipid profile ( total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides in mmol/l). | Assessment will be measured next day after 15th procedure of the IHHT procedure.
  Taken in blood.
Assess the effect of interval hypoxy-hyperoxic training (IHHT) on the trimethylamine n-oxide in mg/dl. | Assessment will be measured next day after 15th procedure of the IHHT procedure.
  Taken in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Yu Kopylov, professor, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- University Clinical Hospital №1 Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Prohibition of local ethics committee

REFERENCES:
- [Derived] Afina AB, Oleg SG, Alexander AB, Ines D, Alexander Yu S, Nikita VV, Denis ST, Daria GG, Zhang Y, Chavdar SP, Dmitriy VG, Elena AS, Irina VK, Philippe Yu K. The Effects of Intermittent Hypoxic-Hyperoxic Exposures on Lipid Profile and Inflammation in Patients With Metabolic Syndrome. Front Cardiovasc Med. 2021 Aug 27;8:700826. doi: 10.3389/fcvm.2021.700826. eCollection 2021. PMID 34513946